CLINICAL TRIAL: NCT00731341
Title: Feasibility Study of Hysteroscopic Cryoablation Treatment of Symptomatic Uterine Fibroids in Women Who do Not Desire Further Pregnancies
Brief Title: Hysteroscopic Cryomyolysis for the Treatment of Submucosal Leiomyomata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFHYS_WH_ 121207 VER 0.1
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Uterine Fibroids; Leiomyoma; Menorrhagia
Keywords: Uterine fibroids; Leiomyoma; Menorrhagia; Hysteroscopic cryoablation; Minimally invasive
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hysteroscopic cryoablation (Experimental): Women undergoing hysteroscopic ultrasound guided cryoablation for the treatment of uterine fibroids.
  Interventions: Procedure: Cryoablation for the treatment of uterine fibroids

INTERVENTIONS:
Procedure: Cryoablation for the treatment of uterine fibroids — Needle will be inserted into the fibroid via the cervix through a hysteroscope channel. Gas is circulated through the sealed needle to form an iceball at the tip. After insertion, the needle will be cooled to a temperature of below -100°C to freeze the tissue of the fibroid.
  Other Names: Presice Cryoablation System; 17-gauge IceBulb™ needle Lot G3021

SUMMARY:
The purpose of the current study is to evaluate the technical success, safety and procedure feasibility of hysteroscopic cryoablation treatment of symptomatic uterine fibroids in women who do not desire further pregnancies using Galil Medical's 17-gauge 400mm Argon-based cryoablation needles

DETAILED DESCRIPTION:
Currently there are no optimal methods for treating symptomatic uterine fibroids. Existing therapeutic options are conservative (medications), invasive (e.g., hysterectomy, surgical myomectomy), or minimally invasive (uterine artery embolization, or myolysis).

Fibroid ablation using cryogenic energy, known as Cryoablation, offers a potential alternative method of fibroid treatment. Cryotherapy is a well-established technique for the treatment of various benign and malignant conditions. Cryoablation has been described for the treatment of prostate cancer, renal cell carcinoma, liver tumors and benign and malignant breast tumors.

Galil Medical's proposed feasibility study is looking to examine the technical success, safety and feasibility of a hysteroscopic approach for the treatment of symptomatic fibroids. This technique involves the insertion and placement of Galil Medical's 17-gauge cryoablation needle(s)guided by a hysteroscopic device. Ultrasound provides real-time monitoring of the needle insertion, placement and iceball propagation during the cryoablation procedure.

This treatment offers the patient to preserve her uterus by a minimally invasive procedure. The type of the fibroids intended for treatment (Type II submucous myomas)are often very difficult to completely and safely remove hysteroscopically and are often treated through an open or laparoscopic procedure. A hysteroscopic procedure does not involve intraperitoneal intervention and is therefore expected to be associated with less intra-operative and post-operative complications.

The recovery from hysteroscopic cryoablation is expected to be fast with only minimal self resolving discomfort. The patient should be able to return to her normal activity within 24-48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Primary complaint is excessive bleeding
* Subject is able to understand and give informed consent for participation in the study
* Pre-menopausal woman between the ages of 30 and 50 (inclusive)
* Has completed childbearing and not contemplating future fertility
* Has symptomatic uterine fibroids
* Fibroids type, size, location and number

  * 1 submucosal fibroid
  * Type I and Type II fibroids
  * 2 to 4cm
* Using contraception to prevent pregnancy

Exclusion Criteria:

* Any evidence of known or suspected infection or pre-malignancy/malignancy
* Desire for future child bearing
* Fibroids

  * Size > 4cm
  * 2 or more submucosal fibroids
  * Fibroid distance from the serosa is less than 1 cm

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas L Thurkow, Principal Investigator — St.Lucas Andreas Ziekenhuis
Locations (1):
- St.Lucas Andreas Ziekenhuis, Amsterdam, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Cryoablation for the Treatment of Uterine Fibroids: All patients in this feasibility study had ultrasound-guided cryoablation of uterine fibroids
Period: Overall Study
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Safety of the procedure will be assessed by incidence and severity of intra and post procedure related adverse events (AEs)
Time Frame: up to 4 weeks post procedure.
Measure: Number; unit: Participants
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Participants | 1

2. Secondary Outcome: Hysteroscopic Cryoablation Related Pain Will be Measured by Self Reported Pain Severity Visual Analogue Scale (VAS) Completed by the Patient
Description: Hysteroscopic cryoablation related pain will be measured by self reported pain severity Visual Analogue Scale (VAS) from a scale of 1 (no pain) to 10 (very severe pain) completed by the patient
Time Frame: Prior to hospital discharge (less than 24 hours post-procedure)
Measure: Mean (Full Range); unit: Units on a scale from 1 to 10
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Units on a scale from 1 to 10 | 1.86 [0 to 3.6]

3. Secondary Outcome: Time (in Days) to Return to Normal Activity
Description: The number of days needed to return to normal activity was assessed by the participant and reported to the investigator. The response was documented at follow-up.
Time Frame: 4 weeks post procedure
Measure: Mean (Full Range); unit: Days
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Days | 6 [1 to 14]

4. Secondary Outcome: Number of Participants Discharged on Day of Cryoablation Procedure.
Description: Per the protocol, this outcome intended to report the average duration of post operative hospital stay. However, this measurement was made very generally and was not collected in number of hours, only the dates were collected. The only actual data that can be stated is that all subjects were discharged from the hospital on the same day as the procedure. In order to report the average length of hospital stay, the wording on the outcome measure title has been changed.
Time Frame: Post procedure
Measure: Number; unit: Participants
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Participants | 3

5. Secondary Outcome: Evaluation of Length of an Average Cryoablation Procedure
Description: Evaluation of length of an average cryoablation procedure for the treatment of uterine fibroids
Time Frame: Post procedure
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Minutes | 65.3 [51 to 74]

6. Secondary Outcome: Physician's Satisfaction From the Ease and Convenience of the Cryoablation Procedure
Description: Physician's satisfaction from the ease and convenience of the cryoablation procedure using a scale of 1 (very satisfied) to 5 (very dissatisfied).
Time Frame: Post procedure
Measure: Mean (Full Range); unit: Score from 1 to 5
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Number analyzed (Participants) | 3
Score from 1 to 5 | 4.3 [4 to 5]

ADVERSE EVENTS:
Time Frame: up to 4 weeks post-procedure
Arm/Group | Cryoablation for the Treatment of Uterine Fibroids
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation for the Treatment of Uterine Fibroids (N=3)
Burning sensation in lower abdomen (Reproductive system and breast disorders) | 1 (1) — This AE occurred in one subject and lasted 6 days before self-resolving. The severity was reported as MILD.

LIMITATIONS AND CAVEATS:
Due to the nature of this feasibility study, a very small number of participants was evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No